CLINICAL TRIAL: NCT05504395
Title: A Phase 1, Single Center, Open Label, Single Dose, Pharmacokinetic and Safety Study of CSTI-500 in Subjects With Prader-Willi Syndrome
Brief Title: A Pharmacokinetic and Safety Study of CSTI-500 in Subjects With Prader-Willi Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ConSynance Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CSTI-500-003
Record Dates: First submitted 2022-08-04; First posted 2022-08-17 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Prader-Willi Syndrome
Keywords: PWS; Phase 1; Single Dose; Non randomized; PK; Safety
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CSTI-500 10mg (Experimental): All eligible subjects will be administered a single oral dose of CSTI-500 10 mg at Visit 2
  Interventions: Drug: CSTI-500

INTERVENTIONS:
Drug: CSTI-500 — Single 10 mg capsule
  Other Names: AMR-001181

SUMMARY:
The purpose of this Phase 1 study is to evaluate the pharmacokinetics (PK) and safety of a single dose of CSTI-500 10 mg in subjects with Prader-Willi syndrome (PWS) between 13 and 50 years of age with a genetically confirmed diagnosis of PWS.

DETAILED DESCRIPTION:
This is an open-label, single center, Phase 1 study to evaluate the PK and safety of a 10 mg single oral dose of CSTI-500, a triple monoamine reuptake inhibitor (TRI), in patients with genetically confirmed PWS. The study will consist of a Screening Period of up to 1-3 days prior to the Baseline Visit (Visit 2). In addition to the Screening Visit (Visit 1), eligible subjects will attend five in-clinic site visits for PK blood draws and safety assessments over a 6-day period. At Visit 2 all subjects will receive one single oral dose of CSTI-500 10 mg. Approximately 14 patients aged 13 to 50 years who meet all eligibility criteria will receive one single dose of CSTI-500.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects (13-50 years of age at screening) with a documented medical record history of PWS confirmed by genetic testing.
* Subject must have a reliable caregiver/parent to bring the subject to the site for the visits, remain with the subject during visit times when allowed to be with the subject and respond to any questions during the visits.
* Female subjects must not be pregnant or lactating and be willing to use double barrier birth control method throughout the study.
* A normal supine systolic blood pressure must be ≤140 mmHg and ≥100 mmHg; diastolic blood pressure must be ≤80 mmHg and ≥60 mmHg at Screening. Pulse rate must be ≥50 bpm and ≤100 bpm and pulse rate increase on standing must be within acceptable range.
* All concomitant medications including blood pressure medications and type 2 diabetic medications must be stable for ≥3 months prior to screening (≤10% change). Supplements and vitamins are not considered concomitant medications for eligibility purposes.

Exclusion Criteria:

* Participation in any clinical study with an investigational drug/device within 3 months prior to screening or during the study.
* Recent use (within 3 months) of weight loss agents including prescription, herbal medications, and weight loss supplements.
* Major surgery within 6 months of screening or planned during the study or history of bariatric surgery.
* Any malignancy in the 2 years prior to screening (excluding basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ that have been successfully treated).
* Current liver, pulmonary, cardiac, or GI disease that would be expected to adversely affect study participation. Stable disease, e.g., asthma or controlled hypertension is not excluded. Liver disease or liver injury as indicated by abnormal liver function tests, ALT, AST, alkaline phosphatase, or serum bilirubin (≥3X ULN for any of these tests).
* Unexplained history or presence of combination of unexplained symptoms e.g., dizziness, syncope, fatigue, palpitations/tachycardia, headaches, or exercise intolerance.
* Heart failure classified per the New York Heart Association (NYHA) level II or greater.
* Myocardial infarction, stroke, or confirmed TIA within the last 5 years.
* Uncontrolled Type 2 diabetes as defined by HbA1c ≥ 9% at Screening.
* Insulin-dependent Type 1 diabetes.
* Subjects with a history of any suicidal behavior.
* Inability to swallow the oral capsule whole with water.

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Pre-dose to 1, 2, 4, 8, 12, 24, 48, 72, and 144 hours post-dose
  Maximum observed plasma concentration following drug administration determined directly from the concentration-time profile.
AUC0-72 | Pre-dose to 1, 2, 4, 8, 12, 24, 48, and 72 hours post-dose
  Area under the plasma-drug concentration-time curve from pre-dose (time 0) to 72 hours after drug administration
AUC0-inf | Pre-dose to 1, 2, 4, 8, 12, 24, 48, 72, and 144 hours post-dose
  Area under the plasma-drug concentration-time curve from pre-dose (time 0) extrapolated to infinite time
CSTI-500 plasma concentration | 1 hour post-dose
CSTI-500 plasma concentration | 2 hour post-dose
CSTI-500 plasma concentration | 4 hour post-dose
CSTI-500 plasma concentration | 8 hour post-dose
CSTI-500 plasma concentration | 12 hour post-dose
CSTI-500 plasma concentration | 24 hour post-dose
CSTI-500 plasma concentration | 48 hour post-dose
CSTI-500 plasma concentration | 72 hour post-dose
CSTI-500 plasma concentration | 144 hour post-dose

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From pre-dose to 15 days post-dose
  Number of participants with TEAEs, defined as an adverse event (AE) that is new or worsened in severity after the dose of study drug. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized by system organ class, preferred term, and treatment.
Incidence of clinically significant findings in physical examinations | Screening to 12, 24, 48, 72, and 144 hours post-dose
Incidence of clinically significant findings in vital signs | Screening and pre-dose to 1, 2, 4, 8, 12, 24, 48, 72, and 144 hours post-dose
  Participants will be assessed for any clinically significant changes in vital parameters (blood pressure, heart rate in supine and standing position, respiratory rate, and body temperature). This also includes evaluation of postural orthostatic tachycardic syndrome.
Incidence of clinically significant findings in laboratory values | Screening to 24, 48, 72, and 144 hours post-dose
  Laboratory evaluations include hematology, thyroid function, and chemistry blood and urine laboratory tests.
Incidence of clinically significant findings in 12-lead electrocardiograms (ECGs) | Screening and pre-dose to 2, 4, 8, 12, 24, 48, 72, and 144 hours post-dose
Comparison of CSTI-500 Cmax values obtained from venous blood draws with values obtained from finger prick samples in PWS subjects | Pre-dose to 1, 2, 4, 8, 12, 24, 48, 72, and 144 hours post-dose
Comparison of CSTI-500 AUC0-72 values obtained from venous blood draws with values obtained from finger prick samples in PWS subjects | Pre-dose to 1, 2, 4, 8, 12, 24, 48, and 72 hours post-dose
Comparison of CSTI-500 AUC0-inf values obtained from venous blood draws with values obtained from finger prick samples in PWS subjects | Pre-dose to 1, 2, 4, 8, 12, 24, 48, 72, and 144 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt Autonomic Dysfunction Center, Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No